CLINICAL TRIAL: NCT00190203
Title: Decompressive Craniectomy In Malignant Middle Cerebral Artery Infarcts : A Sequential Design, Multicenter, Randomized, Controlled Trial
Brief Title: Decompressive Craniectomy In Malignant Middle Cerebral Artery Infarcts
Acronym: DECIMAL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: the study is publiched
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Amel Ouslimany, Department Clinical Research of Departement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P001004; AOM00148
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2008-01-17 (Estimated); Status verified 2007-09

CONDITIONS: Malignant Middle Cerebral Artery Infarction
Keywords: Malignant middle cerebral artery infarction; Decompressive surgery; Hemicraniectomy; Brain edema
MeSH Terms: conditions — Brain Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): HEMICRANIECTOMY
  Interventions: Procedure: Decompressive hemicraniectomy and duraplasty; Procedure: hemicraniectomy

INTERVENTIONS:
Procedure: Decompressive hemicraniectomy and duraplasty — Decompressive hemicraniectomy and duraplasty
Procedure: hemicraniectomy — hemicraniectomy

SUMMARY:
The purpose of this study is to determine if patients with malignant middle cerebral artery infarction have a better clinical outcome after early decompressive surgery compared to standard medical management.

DETAILED DESCRIPTION:
The Decompressive Craniectomy In MALignant middle cerebral artery infarction (DECIMAL) trial is a prospective, multicenter, randomized, open (single blind for the evaluation of the primary outcome measure) controlled study of the efficacy of decompressive craniectomy plus the standard medical therapy as compared with the standard medical therapy alone in patients with a malignant middle cerebral artery infarction. The study protocol is approved by a regional ethic committee (CCPPRB Hospital SAINT LOUIS, PARIS). The study is conducted in 13 stroke centers in France and is funded by the French Ministry of Health and the "ASSISTANCE PUBLIQUE- HOPITAUX DE PARIS". An independent Data Safety Monitoring Board (DSMB) monitors the safety, progress and ethics of the trial.

The aim of the trial is to determine if patients with malignant middle cerebral artery infarction have a better clinical outcome after early decompressive surgery compared to standard medical therapy alone.

Secondary objectives are to determine clinical or MRI based prognostic factors of better outcome after decompressive surgery.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and CT scan signs of complete infarction of the middle cerebral artery
* Onset of symptoms < 30 hours to a possible surgical intervention (< 24 hours for the inclusion and possibility to start treatment/surgery within 6 hours after randomisation)
* DWI infarct volume > 145 cm3

Exclusion criteria:

* The patients having a neurological pre existing handicap (score of Rankin sup or equal in 2).
* Patients having an ischaemia lateral against significant.
* Patients having a haemorrhagic transformation(conversion) sup in 50 % of the territory of the infarct.
* Patients having a severe co-morbidity with a reduced life expectation.
* Patients having a severe cardio-respiratory co-morbidity.
* Patients having antecedent of DUROPLASTIE with transplant of dura mater or transplant of cornea.
* Patients having a thrombolyses in 24 last hours.
* Patients having a severe coagulopathies.
* Patients having one against indication in the general anesthetic.
* Patients for whom a medical follow-up is not possible.
* The pregnant women.
* The patients to whom the surgical operation cannot be realized within 6 hours following the randomisation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2001-12; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Primary endpoint: Functional outcome at 6 months | at 6 months

SECONDARY OUTCOMES:
Secondary endpoints: | during the study
Mortality | during the study
Functional outcome at 9 and 12 months (mRS, NIHSS, Barthel-index) after stroke | at 9 and 12 months and after stroke
Quality of life at 6 and 12 months (SIS) | at 6 and 12 months
Complications related to surgery | during the study
Infarct size at day 5-14 and week 12 and 48 | at day 5-14 and week 12 and 48
Brainstem lesions on T2* after day 5-14 and week 12 and 48 | after day 5-14 and week 12 and 48

CONTACTS AND LOCATIONS:
Overall Officials: Katayoun VAHEDI, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Lariboisière, Assistance Publique - Hôpitaux de Paris, Paris, France

REFERENCES:
- [Result] Vahedi K, Hofmeijer J, Juettler E, Vicaut E, George B, Algra A, Amelink GJ, Schmiedeck P, Schwab S, Rothwell PM, Bousser MG, van der Worp HB, Hacke W; DECIMAL, DESTINY, and HAMLET investigators. Early decompressive surgery in malignant infarction of the middle cerebral artery: a pooled analysis of three randomised controlled trials. Lancet Neurol. 2007 Mar;6(3):215-22. doi: 10.1016/S1474-4422(07)70036-4. PMID 17303527